CLINICAL TRIAL: NCT06206044
Title: Predicting Spinal Failure With Blunt Needle Pinprick Sensory Testing
Brief Title: Evaluation of the Typical Spinal Block During Cesarean Delivery
Status: Enrolling by invitation | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Brandon M Togioka, Principal Investigator, Oregon Health and Science University
Other Study IDs: 25364
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Cesarean Section; Anesthesia, Obstetric
Keywords: Spinal anesthesia; bupivacaine; Sensory dermatomal level
MeSH Terms: interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Study Cohort: Healthy pregnant women of BMI between 20 and 40 kg/m2, height between 5 feet 2 inches and 5 feet 10 inches, who are having cesarean delivery under spinal or combined spinal epidural anesthesia.
  Interventions: Drug: Intrathecal 1.6 ml 0.75% bupivacaine in 8.25% dextrose combined with 15 mcg fentanyl and 150 mcg preservative-free morphine

INTERVENTIONS:
Drug: Intrathecal 1.6 ml 0.75% bupivacaine in 8.25% dextrose combined with 15 mcg fentanyl and 150 mcg preservative-free morphine — Patients will receive standard intrathecal medications for urgent and scheduled cesarean delivery at the study site. All study subjects will receive bupivacaine, fentanyl, and morphine.
  Other Names: Marcaine

SUMMARY:
This will be a prospective, observational, single-center study to evaluate the accuracy of sensory testing by blunt 16-gauge plastic cannula during the 15 minutes after spinal injection for predicting spinal failure. While previous studies assessed the minimal sensory level required for painless cesarean delivery at skin incision or delivery, no studies have assessed the accuracy of sensory testing at an earlier time point.

DETAILED DESCRIPTION:
Primary Objective:

1. Evaluate the accuracy of sensory testing with blunt plastic 16-gauge cannula during the 15 minutes after spinal injection for predicting spinal failure. Cephalad sensory dermatomal levels will be assessed at 1 (t1), 3 (t3), 5 (t5), 7 (t7), 9 (t9), 11 (t11), 13 (t13), and 15 (t15) minutes after intrathecal 1.6 ml 0.75% bupivacaine in 8.25% dextrose combined with 15 mcg fentanyl and 150 mcg morphine (study solution). Spinal failure, which is defined as inability to achieve a T4 level to pinprick by the 15-minute timepoint or intraoperative pain (VAS > 0) requiring treatment

Secondary Objectives:

1. Conversion to another anesthetic technique (general anesthesia or activation of the epidural catheter)
2. Inadequate anesthesia (analgesic supplementation with ketamine, > 20 mg propofol, > 2 mg midazolam, > 10 mg parental morphine equivalents, or intraperitoneal chloroprocaine).
3. Patient satisfaction upon arrival to the postanesthesia care unit, rated on a 1-5 Likert scale

A sample size calculation

Population: 250 pregnant females undergoing non-emergency cesarean section delivery in the Labor & Delivery Operating Rooms at Oregon Health & Science University.

Number of Sites: Single center trial

Study Duration: Institutional Review Board approval has been obtained. Study initiation, enrollment, and data collection is expected to take 24 months. Data analysis, manuscript writing, editing, submission and revision to a peer-reviewed journal is expected to take an additional 6 months.

In summary, the study should be completed in under 3 years.

Subject Participation Duration: Total time of subject participation including time for recruitment, enrollment, data collection during the preanesthesia consult, and post-consult data collection will be less than 3 hours.

Estimated Time to Complete Enrollment: Estimated time from enrollment into study of the first subject to enrollment into study of the last subject is 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cesarean delivery under spinal or combined spinal epidural anesthesia
* BMI between 20 and 40 kg/m2
* Height between 5 feet 2 inches and 5 feet 10 inches.
* English and non-English speaking patients, if interpretive services are available

Exclusion Criteria:

* Patient refusal
* Contraindications to neuraxial anesthesia (coagulopathy, CNS pathology, infection at site of needle puncture)
* Allergy to any study medications
* Use of epidural anesthesia
* Emergency (red) cesarean delivery
* Conditions that impact dermatomal sensory testing including spinal cord injury with sensory deficits and abdominoplasty
* Prison inmates
* Decisionally impaired individuals
* Pregnancies involving multiple fetuses

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Participants must be biologically female, this study evaluates spinal anesthesia given to pregnant individuals undergoing cesarean section delivery
Study Population: Pregnant females receiving spinal or combined spinal epidural anesthesia for cesarean delivery
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with spinal failure | 90 minutes
  A composite outcome that will be categorized as "yes" if there is either preoperative or intraoperative spinal failure. Preoperative failure will be defined as failure to achieve a T4 level to pinprick by the 15-minute timepoint. Intraoperative failure will be defined as pain (VAS > 0) that requires anesthesia provider medication administration.
  Pain will be queried at time of skin incision, fetal delivery, uterine exteriorization, uterine interiorization or end of uterine closure, and end of skin closure. If VAS > 0, the anesthesia provider will ask the patient if they would like analgesic medication.
  Discomfort at any other time during the cesarean delivery that is treated with neuraxial or intravenous analgesia will also count.
  Pain will be rated according to the scale: 0 = no pain, 10 = worst pain imaginable

SECONDARY OUTCOMES:
Number of participants with conversion to another anesthetic technique | 90 minutes
  Conversion to general anesthesia or activation of the epidural catheter for intraoperative pain
Number of participants with inadequate anesthesia | 90 minutes
  Analgesic supplementation with ketamine, > 20 mg propofol, > 2 mg midazolam, > 10 mg parental morphine equivalents, or intraperitoneal chloroprocaine
Patient satisfaction assessed by 5-point Likert scale, minimum value=1, maximum value=5, with higher values representing better patient satisfaction | 2 Hours
  Patient satisfaction upon arrival to the post-anesthesia care unit, rated on a 1-5 Likert scale with higher values representing better patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M Togioka, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Due to patient data protection regulations within the study site there is not a plan to make individual participant data available to other researchers. Reasonable requests emailed to the PI will considered on a case-by-case basis.

REFERENCES:
- [Background] Kinsella SM. A prospective audit of regional anaesthesia failure in 5080 Caesarean sections. Anaesthesia. 2008 Aug;63(8):822-32. doi: 10.1111/j.1365-2044.2008.05499.x. Epub 2008 Jun 28. PMID 18547291
- [Background] Russell IF. A comparison of cold, pinprick and touch for assessing the level of spinal block at caesarean section. Int J Obstet Anesth. 2004 Jul;13(3):146-52. doi: 10.1016/j.ijoa.2003.12.007. PMID 15321392
- [Background] Ousley R, Egan C, Dowling K, Cyna AM. Assessment of block height for satisfactory spinal anaesthesia for caesarean section. Anaesthesia. 2012 Dec;67(12):1356-63. doi: 10.1111/anae.12034. Epub 2012 Oct 12. PMID 23061397
- [Background] Hoyle J, Yentis SM. Assessing the height of block for caesarean section over the past three decades: trends from the literature. Anaesthesia. 2015 Apr;70(4):421-8. doi: 10.1111/anae.12927. Epub 2014 Nov 10. PMID 25388969
- [Background] Russell IF. Levels of anaesthesia and intraoperative pain at caesarean section under regional block. Int J Obstet Anesth. 1995 Apr;4(2):71-7. doi: 10.1016/0959-289x(95)82995-m. PMID 15636981
- [Background] de Souza Soares EC, Balki M, Downey K, Ye XY, Carvalho JCA. Assessment of sensory block during labour epidural analgesia: a prospective cohort study to determine the influence of the direction of testing. Can J Anaesth. 2022 Jun;69(6):750-755. doi: 10.1007/s12630-022-02228-x. Epub 2022 Mar 14. PMID 35289377
- [Background] Yentis SM. Height of confusion: assessing regional blocks before caesarean section. Int J Obstet Anesth. 2006 Jan;15(1):2-6. doi: 10.1016/j.ijoa.2005.06.010. Epub 2005 Oct 26. No abstract available. PMID 16256334

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT06206044/Prot_SAP_000.pdf